CLINICAL TRIAL: NCT01863706
Title: Safety and Efficacy of Misoprostol Versus Oxytocin for Prevention of Post Partum Hemorrhage
Brief Title: Misoprostol Versus Oxytocin for Prevention of Post Partum Hemorrhage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Mahboobi, Dr, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Misoprostol for PPH
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Post Partum Hemorrhage
Keywords: Misoprostol; Oxytocin; Post Partum Hemorrhage (PPH); Third stage of labour
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): 400µg oral misoprostol
  Interventions: Drug: Misoprostol
- Oxytocin (Active Comparator): 20 IU oxytocin
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — 400µg oral misoprostol
  Other Names: Cytotec
  Arms: Misoprostol
Drug: Oxytocin — 20 IU Oxytocin
  Other Names: Syntocinon
  Arms: Oxytocin

SUMMARY:
Post partum Hemorrhage (PPH) is one of three main causes of death in pregnant women. Oxytocin is widely used for prevention of PPH. Some studies suggested misoprostol as an alternative treatment when Oxytocin isn't available. The aim of this study is to compare the safety and efficacy of Oxytocin and misoprostol for prevention of PPH.

DETAILED DESCRIPTION:
In a double blind randomized controlled trial 400 pregnant women who has vaginal delivery at Shariati hospital are assigned into two groups either to receive 20 unite oxytocin in 1000cc ringer and 2 placebo tablet or 400mcg oral misoprostol and 2cc normal saline in 1000cc ringer.

ELIGIBILITY:
Inclusion Criteria:

* were women with singleton pregnancy
* with cephalic presentation
* who had NVD spontaneously or by induction

Exclusion Criteria:

* placenta previa
* placental detachment
* coagulation problems
* previous CS
* macrosomia
* Polyhydramnios
* and uncontrolled asthma

Ages: 10 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Amount of bleeding | 1 hour
  within 1 hours after delivery

SECONDARY OUTCOMES:
Hemoglobin decrease | 24 hours
Hematocrite decrease | 24 hours

OTHER OUTCOMES:
Side effects | 24 hours
  Diarrhea, Vommiting, Fever, Chills

CONTACTS AND LOCATIONS:
Overall Officials: Minoo Rajaei, Dr, Study Chair — Hormozgan University of Medical Sciences; Zohreh Shahboodaghi, Dr, Study Director — Hormozgan University of Medical Sciences
Locations (1):
- Hormozgan University of Medical Sciences, Bandar Abbas, Hormozgan, Iran

REFERENCES:
- [Derived] Rajaei M, Karimi S, Shahboodaghi Z, Mahboobi H, Khorgoei T, Rajaei F. Safety and efficacy of misoprostol versus oxytocin for the prevention of postpartum hemorrhage. J Pregnancy. 2014;2014:713879. doi: 10.1155/2014/713879. Epub 2014 Mar 5. PMID 24734184